CLINICAL TRIAL: NCT03715790
Title: Improve Sudden Cardiac Arrest (SCA) Bridge Study
Brief Title: Improve SCA Bridge Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT18019
Record Dates: First submitted 2018-10-03; First posted 2018-10-23 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2023-04

CONDITIONS: Sudden Cardiac Arrest; Acute Myocardial Infarction
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EP Referred Group: Subjects with EF ≤ 40% or meeting one of the referral criteria
  Interventions: Behavioral: EP referred group
- Non-Referred Group: Subjects with 40%< EF <50%.
  Interventions: Behavioral: Non-Referred group

INTERVENTIONS:
Behavioral: EP referred group — Referred for sudden cardiac death (SCD) risk stratification and management
  Groups: EP Referred Group
Behavioral: Non-Referred group — Not referred for sudden cardiac death (SCD) risk stratification and management.
  Groups: Non-Referred Group

SUMMARY:
The purpose of the Improve SCA Bridge study is to characterize the care pathway flow of post-acute myocardial infarction (MI) patients as a result of standard assessments of left ventricular ejection fraction (LVEF) in the acute phase (≤14 days post- acute MI) and chronic phase (≥40-90 days post-acute MI).

DETAILED DESCRIPTION:
To determine how many patients are referred for sudden cardiac death (SCD) risk stratification and management, indicated for implantable cardioverter defibrillator (ICD), or cardiac resynchronization therapy- defibrillator (CRT-D) implant, and how many receive such devices within 12 months of experiencing an MI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above (or meet age requirements per local law)
* Patients who have an acute Myocardial Infarction (MI) (STEMI or Non-STEMI) ≤ 30 days of study enrollment and have a LVEF <50% measurement ≤ 14 days post-acute MI
* Willing and able to give valid Informed Consent

Exclusion Criteria:

* Patient has previously received or currently implanted with an ICD or CRT-D
* Patient has any contraindication for ICD/CRT-D
* Patient has a life expectancy of less than 12 months
* Patient who has had an EP referral within the last 12 months
* Any exclusion criteria required by local law (e.g. pregnancy, breast feeding etc.)
* Patient is unable (e.g. mental disorder) or unwilling to be compliant with the responsibilities as specified in the informed consent form.
* Patient is enrolled in a concurrent study that has not been approved for concurrent enrollment by the Medtronic Clinical Trial Leader

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have an acute Myocardial Infarction (MI) (STEMI or Non-STEMI).
Sampling Method: Probability Sample
Enrollment: 1491 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu Zhang, Principal Investigator — Fuwai Hospital Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (52):
- National Heart Foundation Hospital and Research Institute, Dhaka, Bangladesh
- Gleneagles Jerudong Park Medical Centre, Brunei, Brunei
- China (15):
  - Fuwai Hospital Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - Peking University First Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chendu
  - Sun Yat-SEN Memorial hospital, Sun Yat-sen University, Guangzhou
  - Guizhou Provincial People's Hospital, Guizhou
  - Hangzhou First People Hospital, Hangzhou
  - Sir Run Run Shaw Hospital School of Medicine Zhejiang University, Hangzhou
  - The first Hospital of Lanzhou Hospital, Lanzhou
  - Nanjing First Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Sichuan Provincial People's Hospital, Sichuan
  - Wuhan Asia heart hospital, Wuhan
  - Xiamen Cardiovascular Hospital, Xiamen
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang
- International Cardic Center, Alexandria, Egypt
- India (5):
  - The Madras Medical Mission, Chennai
  - Eternal Hospital, Jaipur
  - Kasturba Medical College Hospital, Mangalore
  - Batra Hospital and Medical Research Centre (BHMRC), New Delhi
  - Fortis Escorts Heart Institute, New Delhi
- Indonesia (2):
  - National Cardiovascular Center Harapan Kita, Jakarta
  - Rumah Sakit Cipto Mangunkusumo, Jakarta
- Malaysia (3):
  - Hospital Serdang, Kajang
  - Queen Elizabeth II Hospital, Kota Kinabalu
  - Sarawak Heart Centre, Kota Samarahan
- National Institute of Cardiovascular Diseases, Karachi, Pakistan
- Chinese General Hospital and Medical Center, Manila, Philippines
- Saudi Arabia (2):
  - King Fahad Armed Forces Hospital, Jeddah
  - Prince Sultan Cardiac Center, Riyadh
- Changi General Hospital, Singapore, Singapore
- South Africa (2):
  - Mediclinic Panorama, Cape Town
  - Netcare Unitas Hospital, Pretoria
- South Korea (9):
  - Chonnam National University Hospital, Gwangju
  - Sejong General Hospital, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Keimyung University Dongsan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital of CGMF, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand
- The Military Hospital of Tunis, Montfleury, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chew DS, Wilton SB, Kavanagh K, Southern DA, Tan-Mesiatowsky LE, Exner DV; APPROACH Investigators. Left ventricular ejection fraction reassessment post-myocardial infarction: Current clinical practice and determinants of adverse remodeling. Am Heart J. 2018 Apr;198:91-96. doi: 10.1016/j.ahj.2017.11.014. Epub 2017 Dec 5. PMID 29653653
- [Result] Adabag AS, Therneau TM, Gersh BJ, Weston SA, Roger VL. Sudden death after myocardial infarction. JAMA. 2008 Nov 5;300(17):2022-9. doi: 10.1001/jama.2008.553. PMID 18984889
- [Result] Chia YMF, Teng TK, Tan ESJ, Tay WT, Richards AM, Chin CWL, Shimizu W, Park SW, Hung CL, Ling LH, Ngarmukos T, Omar R, Siswanto BB, Narasimhan C, Reyes EB, Yu CM, Anand I, MacDonald MR, Yap J, Zhang S, Finkelstein EA, Lam CSP. Disparity Between Indications for and Utilization of Implantable Cardioverter Defibrillators in Asian Patients With Heart Failure. Circ Cardiovasc Qual Outcomes. 2017 Nov;10(11):e003651. doi: 10.1161/CIRCOUTCOMES.116.003651. PMID 29150533
- [Result] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines; American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines: developed in collaboration with the American College of Emergency Physicians and Society for Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2013 Jul 1;82(1):E1-27. doi: 10.1002/ccd.24776. Epub 2013 Jan 8. No abstract available. PMID 23299937
- [Derived] Zhang S, Chen WJ, Sankardas MA, Ahmed WH, Liew HB, Gwon HC, Nesa Malik FT, Tang B, Haggui A, Oh IY, Ong TK, Cheng CI, Liu X, Seth A, Choi YJ, Qamar N, Rungpradubvong V, Wang CC, Jeon J, Wong G, Lemme F, Van Dorn B, Lexcen D, Huang D; Improve Sudden Cardiac Arrest Bridge Investigators. Improve the Prevention of Sudden Cardiac Arrest in Patients With Post-Acute Myocardial Infarction. JACC Asia. 2022 Sep 20;2(5):559-571. doi: 10.1016/j.jacasi.2022.06.006. eCollection 2022 Oct. PMID 36518723

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While the study objective was to categorize patients into those who met referral criteria and those who did not, those two groups were not, strictly speaking, considered to be treatment arms. Rather, subjects in the single enrolled patients arm could, by meeting the required criteria at any of the three follow-up evaluations, be reported in the referral group. Thus the two groups were the result of the collective referral assessments and not separate study arms with a subsequent study flow.
Groups:
- Post-acute MI Patients Who Are Candidates for SCA Risk Stratification: Subjects who were enrolled in the Improve SCA Bridge Study and were not excluded due to not meeting inclusion/exclusion criteria
Period: 3-months
Arm/Group | Post-acute MI Patients Who Are Candidates for SCA Risk Stratification
Started | 1491
Completed | 1170
Not Completed | 321
Period: 6-months
Arm/Group | Post-acute MI Patients Who Are Candidates for SCA Risk Stratification
Started | 1170
Completed | 916
Not Completed | 254
Period: 12-months
Arm/Group | Post-acute MI Patients Who Are Candidates for SCA Risk Stratification
Started | 916
Completed | 887
Not Completed | 29

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Subjects: Subjects who were enrolled in the Improve SCA Bridge Study and were not excluded due to not meeting inclusion/exclusion criteria
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 1491
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263
  Male | 1228
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Singapore | 19
  Philippines | 1
  Egypt | 15
  Malaysia | 86
  Thailand | 22
  India | 267
  Saudi Arabia | 70
  Brunei | 30
  Bangladesh | 80
  South Korea | 237
  Pakistan | 50
  China | 394
  Taiwan | 120
  South Africa | 12
  Tunisia | 50
  Indonesia | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Post-Acute MI Patients Who Are Referred for Sudden Cardiac Death Risk Stratification > Risk (SCD) Stratification and Management
Description: The numerator for this endpoint will be defined as the number of patients who met the clinician's determination to refer the subject for SCD risk stratification and management at any of the three follow-up visits. The denominator for this endpoint is the number of patients who completed a 3-month follow-up visit. While the participant study flow is composed of "referred" and "not referred" groups, these groups are simply the results of the referral process in the single arm of enrolled patients. Thus the analysis of the endpoints is conducted within this one arm.
  No hypotheses were tested for this endpoint.
Time Frame: 3-months post-MI to 12-months post-MI
Population: Enrolled subjects who were evaluated at 3-month follow up to determine if they met referral criteria or did not meet referral criteria.
Measure: Count of Participants; unit: Participants
Groups:
- Referred Subjects: Subjects who were referred for SCA risk stratification
- Not Referred Subjects: Subjects who were not referred for SCA risk stratification
Arm/Group | Referred Subjects | Not Referred Subjects
Number analyzed (Participants) | 1170 | 1170
Participants | 236 | 934

2. Secondary Outcome: Percentage of Post-Acute MI Patients Who Are Known to be Indicated for an ICD/CRT-D Within 12 Months Post-MI
Description: The numerator for this endpoint will be the number of subjects who were indicated for an ICD/CRT-D device during any of the three follow-up visits. The denominator will be the number of subjects who completed a 3-month follow-up visit.
  While the participant study flow is composed of "referred" and "not referred" groups, these groups are simply the results of the referral process in the single arm of enrolled patients. Thus the analysis of the endpoints is conducted within this single arm. The analysis cannot be performed within the "referred" and "not referred" groups as patients not referred are not eligible for the secondary endpoints involving device indication or implant.
  No hypotheses were tested for this endpoint.
Time Frame: 3-months post-MI to 12-months post-MI
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Post-acute MI Subjects: Subjects that were enrolled in the Improve SCA Bridge study that were not excluded due to not meeting inclusion/exclusion criteria AND attended a follow-up visit
Arm/Group | Post-acute MI Subjects
Number analyzed (Participants) | 1170
Participants | 127

3. Secondary Outcome: Percentage of Post-Acute MI Patients Who Receive an ICD/CRT-D Within 12 Months Post-MI.
Description: The numerator for this endpoint will be the number of subjects who received an ICD/CRT-D device during any of the three follow-up visits. The denominator for this endpoint will be the number of patients who completed a 3-month follow-up visit.
  While the participant study flow is composed of "referred" and "not referred" groups, these groups are simply the results of the referral process in the single arm of enrolled patients. Thus the analysis of the endpoints is conducted within this single arm. The analysis cannot be performed within the "referred" and "not referred" groups as patients not referred are not eligible for the secondary endpoints involving device indication or implant.
  No hypotheses were tested for this endpoint.
Time Frame: 3-months post-MI to 12-months post-MI
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-acute MI Subjects
Number analyzed (Participants) | 1170
Participants | 18

4. Secondary Outcome: Percentage of ICD Indicated Patients Who Were Not Referred, Refused Referral or Refused Implant of an ICD
Description: The outcome measure will be the percentage of patients with ICD indication, who were not referred, refused referral or refused implant. The denominator will count all patients with at least one of the below:
  1. a reduced ejection fraction, as measured by the Left Ventricular Ejection Fraction (LVEF) being lower or equal than 40%.
     >
  2. ventricular arrhythmia, AV block, new onset bundle branch block, or conduction abnormalities as measured by ECGs.
     >
  3. unexplained syncope, clinically significant palpitations or symptomatic bradycardia as assessed by the physician.
     > The numerator will count the patients included in the denominator who were not referred, refused referral or refused implant of an ICD/CRT-D.
     While the participant study flow is composed of "referred" and "not referred" groups, these groups are simply the referral process results in the single arm of enrolled patients, with analysis performed within this arm.
     No hypotheses were tested for this endpoint.
Time Frame: 3-months post-MI to 12-months post-MI
Population: Enrolled patients who, at the 3-month visit, met the criteria for referral for SCD risk stratification. These criteria include a reduced ejection fraction less than or equal to 40%, ventricular arrhythmia, AV block, new onset bundle branch block, or conduction abnormalities, or unexplained syncope, clinically significant palpitations or symptomatic bradycardia.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Who Met Referral Criteria: All patients indicated for ICD/CRT-D with at least one of the below:
  1. a reduced ejection fraction, as measured by the Left Ventricular Ejection Fraction (LVEF) being lower or equal than 40%.
     >
  2. ventricular arrhythmia, AV block, new onset bundle branch block, or conduction abnormalities as measured by ECGs.
     >
  3. unexplained syncope, clinically significant palpitations or symptomatic bradycardia as assessed by the physician.
Arm/Group | Subjects Who Met Referral Criteria
Number analyzed (Participants) | 398
Participants
  Number of patients who who were not referred, refused referral or refused implant of an ICD/CRT-D | 162
  Number of patients not referred due to "the patient deemed referral not necessary". | 21
  Number of patients not referred due to "the patient was asymptomatic". | 42
  Number of patients not referred due to "the physician preferred continuing with medication". | 75
  Number of patients who refused implant due to "patient does not want risk associated with implant". | 40
  Number of patients who refused implant due to "patient does not believe in benefit of ICD/CRT-D". | 36
  Number of patients who refused implant due to "patient unable to pay for device". | 62

5. Secondary Outcome: Percentage of Post-Acute MI Patients Who Experience Cardiovascular Mortality
Description: The numerator for this endpoint will be the number of patients who experience cardiovascular mortality. The denominator will be the number of patients enrolled in the study.
  No hypotheses were tested for this endpoint.
Time Frame: Enrollment to 12-months post-MI
Population: Enrolled subjects
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Subjects: Subjects that were enrolled in the Improve SCA Bridge study that were not excluded due to not meeting inclusion/exclusion criteria.
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 1491
Participants | 29

6. Secondary Outcome: Evolution of the Ejection Fraction Over the Immediate Period of Post MI
Description: The Left Ventricular Ejection Fraction (LVEF) will be measured acutely post MI (≤14 days after MI onset) and chronically (40-90 days). The acute measurement will occur over all 1491 subjects assessed at baseline, while the chronic assessment will be measured over the 1046 subjects with a 3-month LVEF assessment. This outcome will compare the average LVEF, by percent, between these two phases.
  No hypotheses were tested for this endpoint.
Time Frame: Enrollment to 3-months post-MI
Population: Acute LVEF measurements occurred at baseline on 1491 subjects. Chronic LVEF measurements were collected at the 3-month follow up on 1046 subjects (104 subjects were exited before the 3-month follow up, and 341 subjects did not have their LVEF measurement taken at the 3-month follow up).
Measure: Mean (Standard Deviation); unit: Percentage of LV stroke volume
Arm/Group | Enrolled Subjects
Number analyzed (Participants) | 1491
Percentage of LV stroke volume
  Acute | 39.8 (6.8)
  Chronic: number analyzed (Participants) | 1046
  Chronic | 46.3 (10.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected starting at baseline through 12-month follow up.
Description: Only deaths and cardiovascular related adverse events were collected for this study.
Groups:
- Enrolled Subjects: Subjects who were enrolled in the Improve SCA Bridge Study and were not excluded due to not meeting inclusion/exclusion criteria.
  While enrolled patients were separated into "Referred" and "Not-Referred" groups based on the outcomes at the 3-month visit, these groups are not separate treatment arms. It would be misleading to compare adverse events between these groups as patients not referred due to an LVEF above 50% were subsequently not followed and had relatively little exposure when compared with the referred patients.
Arm/Group | Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 88/1491
Serious Adverse Events (participants affected / at risk) | 180/1491
Other Adverse Events (participants affected / at risk) | 18/1491
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=1491)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 7 (7)
Acute Left Ventricular Failure (Cardiac disorders) | 5 (5)
Acute Myocardial Infarction (Cardiac disorders) | 24 (26)
Angina Pectoris (Cardiac disorders) | 7 (8)
Angina Unstable (Cardiac disorders) | 4 (4)
Arrhythmia (Cardiac disorders) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 7 (7)
Cardiac Failure (Cardiac disorders) | 9 (11)
Cardiac Failure Acute (Cardiac disorders) | 25 (28)
Cardiac Failure Chronic (Cardiac disorders) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 5 (6)
Cardio-Respiratory Arrest (Cardiac disorders) | 4 (4)
Cardiogenic Shock (Cardiac disorders) | 4 (4)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 16 (17)
Intracardiac Thrombus (Cardiac disorders) | 2 (2)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1)
Left Ventricular Failure (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Myocardial Rupture (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 3 (3)
Ventricular Septal Defect Acquired (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Accidental Death (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Death (General disorders) | 22 (22)
Multiple Organ Dysfunction Syndrome (General disorders) | 2 (2)
Sudden Cardiac Death (General disorders) | 13 (13)
Sudden Death (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Cerebellar Infarction (Nervous system disorders) | 1 (1)
Cerebral Infarction (Nervous system disorders) | 2 (2)
Cerebrovascular Accident (Nervous system disorders) | 3 (3)
Embolic Stroke (Nervous system disorders) | 1 (2)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Stenosis (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects (N=1491)
Angina Pectoris (Cardiac disorders) | 6 (6)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1)
Atrioventricular Block (Cardiac disorders) | 1 (1)
Cardiac Aneurysm (Cardiac disorders) | 1 (1)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 4 (4)
Dizziness Postural (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data after release of a multi-center publication per the publication strategy following Medtronic's review for disclosure of confidential information ("CI"), technical correctness, disclosure of patentable or copyrightable material, and selection and order of publications by the publications committee. Any such CI and/or item identified as not technically correct is deleted prior to publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03715790/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT03715790/SAP_001.pdf